CLINICAL TRIAL: NCT06133595
Title: A Multicenter, Waitlist Controlled, Randomized Clinical Trial of the Effectiveness of Mi Bridge, a Motivational Interviewing Intervention to Facilitate Help-seeking Among Individuals with Sexual Interest in Children
Brief Title: Mi Bridge - Motivational Interviewing to Facilitate Help-seeking Among Individuals with Sexual Interest in Children
Acronym: Mi Bridge
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Karolinska Institutet (Other)
Collaborators: Centre for Psychiatry Research, Region Stockholm, Sweden (Unknown); Linkoeping University (Other Government); Universitat Jaume I, Spain (Unknown); Protect Children Organisation, Finland (Unknown); National Institute of Mental Health, Czech Republic (Other); Academy of the Police Force, Bratislava, Slovakia (Unknown); Universitätsklinikum Hamburg-Eppendorf (Other)
Responsible Party: Principal Investigator, Christoffer Rahm, Principal Investigator, Karolinska Institutet
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 2023-02321-01-B; 101084355-BRIDGE-ISF-2021 (Other: European Commission)
Record Dates: First submitted 2023-10-12; First posted 2023-11-15 (Actual); Last update posted 2024-10-10 (Actual); Status verified 2024-10

CONDITIONS: Child Sexual Abuse; Pedophilia
Keywords: Child sexual abuse material; Motivational Interviewing; Evidence based treatment; Individuals with sexual interest in children
MeSH Terms: conditions — Pedophilia

STUDY DESIGN:
Intervention Model Description: Participants are allocated to either the Mi Bridge intervention or waitlist during the initial phase of the study and those who receive waitlist receive Mi Bridge during the second phase of the study.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Experimental: MiBridge (Experimental): MiBridge: A series of five conversations over three weeks to help participants understand more about themselves and their willingness to change, and to help participants connect with the care they need and want.
  Interventions: Behavioral: Behavioral: MiBridge
- No Intervention: Waitlist (No Intervention): Participants are on a waitlist which means they have no active intervention, only weekly measurements with the same questionnaires as in the active arm

INTERVENTIONS:
Behavioral: Behavioral: MiBridge — A series of five conversations over three weeks to help participants understand more about themselves and their willingness to change, and to help participants connect with the care they need and want.
  Arms: Experimental: MiBridge

SUMMARY:
The overall aim of the study is to evaluate the effectiveness of Mi Bridge to motivate high risk participants to admit to treatment.

The main research question is:

Is Mi Bridge, an anonymous online program based on the principles for Motivational Interviewing, effective in making high risk individuals for committing child sexual abuse prone to seek treatment for problems related to sexual interest involving children at a health care facility?

DETAILED DESCRIPTION:
The present research project aims to contribute to the further development of accessible, evidence-based and safe care for people with sexual interest in children, and that are using child sexual abuse material (CSAM), so that these people can access treatment according to their needs and level of risk, with the objective of reducing the risk for child sexual abuse and improving the health of the group.

The intervention will be available in seven languages and will be tested in six countries.

Primary research questions:

Does Mi Bridge increase the likelihood that individuals at high risk for committing child sexual abuse accept seeking treatment for problems related to sexual interest involving minors at a health care facility?

Does Mi Bridge increase participants motivation for change regarding sexual behaviors involving minors?

Secondary research questions:

Does Mi Bridge increase the intention to seek treatment in the coming month for problems related to sexual interest involving minors at a health care facility?

Does Mi Bridge decrease participants sexual interest involving children?

Does Mi Bridge significantly decreases participants past week sexual behaviors involving children?

Does Mi Bridge significantly decreases participants symptoms of depression?

Is Mi Bridge effective in reducing certain dynamic risk factors for committing child sexual abuse?

About the intervention. Mi Bridge is a series of up to five conversations between a practitioner and a study participant over three weeks to help the participants understand more about themselves and their willingness to change, and to help the participants connect with the care they need and want. The conversations are carried out as anonymous voice calls or anonymous text-based chat. Mi Bridge is based on the established and well-researched method of Motivational Interviewing, which has been shown to be effective in helping people achieve the desired changes for several lifestyle related problems.

Research subjects will be recruited through Darknet and Clearnet. Darknet refers to websites that are accessible via Tor or similar services. The intervention is provided by practitioners and researchers in the relevant countries.

Mi Bridge will be evaluated through an international multicenter study using randomized wait-list controlled design.

The research subjects will sign a written consent form on the Iterapi platform without disclosing personal data such as name or location. During the subsequent screening interview via chat or voice call on Iterapi, participation criteria are ensured, questions are answered, and the consent to participate is confirmed. The research subjects are thus admitted to the study.

After inclusion, participants answer the baseline survey which consists of validated self-assessment questionnaires with both multiple choice and free-text answers.

Weekly during, after the waitlist, and after the therapeutic intervention, research subjects answer questions to evaluate the effectiveness and safety of the interventions.

A Statistical Analysis Plan (SAP) based on pilot study is pre-registered at the OSF platform. The SAP describes sample size calculations, and planned analyses of outcome measures.

ELIGIBILITY:
Inclusion Criteria:

* Sufficient language skills: English, Swedish, Finnish, Czech, Slovak, German, or Spanish

  * Concerns about sexual interest regarding children
  * CSAM use past six month
  * High risk for committing child sexual abuse according to the SChiMRA scale

Exclusion Criteria:

* Participants with a severe psychiatric illness (such as high acute suicide risk or severe substance abuse) will be excluded, or lack of serious intentions to participate.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2023-09-18 (Actual); Primary Completion 2024-10-08 (Estimated); Study Completion 2024-10-08 (Estimated)

PRIMARY OUTCOMES:
Motivation to seek treatment | Pre-intervention, during the intervention, and immediately after the intervention.
  The Motivation to Seek Care questionnaire, item 1, which targets motivation to seek treatment for problems related to sexual interest involving children (Likert scale 1-7; higher scores indicates higher motivation).
Motivation to make a change | Pre-intervention, during the intervention, and immediately after the intervention.
  Responses on the Change Questionnaire (3 items, ordinal from 0 - 10; 0 - 30 points in total; higher score indicates more readiness to make a change related to sexual behaviors involving children).

SECONDARY OUTCOMES:
Plan to seek treatment coming month | Pre-intervention, during the intervention, and immediately after the intervention.
  The Motivation to Seek Care questionnaire, item 2, which targets the intention to actually seek treatment during the coming month for problems related to sexual interest involving children (Y/N, coded as 1=YES, and 2=NO).
Sexual interest involving children | Pre-intervention, during the intervention, and immediately after the intervention.
  Measured by Sexual Symptom Assessment Scale (SASS)(0-48 points; higher scores indicate more interest).
Behaviors related to sexual interest in children | Pre-intervention, during the intervention, and immediately after the intervention.
  Time spent last week (hours), as self reported on the SChiMRA+ part B, item 1-4.
Level of hypersexuality | Pre-intervention, during the intervention, and immediately after the intervention.
  Scores on the HBI-19 questionnaire (Hypersexual Behavior Inventory; 19-95 points; higher scores indicate higher level of sexuality; more than 52 points indicate hypersexuality).
Dynamic risk for committing child sexual abuse | Pre-intervention, during the intervention, and immediately after the intervention.
  Scores on Acute-2007 (21 items; 0-42 points; higher scores indicate higher dynamic risk for committing child sexual abuse).
Depressive symtoms | Pre-intervention, during the intervention, and immediately after the intervention.
  Scores on the PHQ-9 questionnaire (Patient Health Questionnaire; 0-27 points; higher scores indicate more severe depressive symptoms).

CONTACTS AND LOCATIONS:
Locations (6):
- National Institute of Mental Health, Klecany, Czechia
- Protect Children NGO, Helsinki, Finland
- University Medical Center Hamburg-Eppendorf, Hamburg, Germany
- Bratislava Police Academy, Bratislava, Slovakia
- Universitat Jaume I, Castellon, Spain
- Centre for psychiatry research, Region Stockholm, Stockholm, Sweden

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Related Info — https://www.iterapi.se/sites/bridge